CLINICAL TRIAL: NCT07177495
Title: Radiographic and Histomorphometric Assessment for Maxillary Sinus Floor Elevation and Augmentation Using A Mixture of 1:1 Autogenous Bone With Deproteinized Bovine Bone Particulate Versus Deproteinized Bovine Bone Particulate: A Randomized Clinical Trial
Brief Title: Radiographic and Histomorphometric Assessment for Maxillary Sinus Floor Elevation and Augmentation Using A Mixture of 1:1 Autogenous Bone With Deproteinized Bovine Bone Particulate Versus Deproteinized Bovine Bone Particulate
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, merna hamdy, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: maxillary sinus lift
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Maxillary Sinus Lifting
Keywords: maxillary sinus lifting; deproteinized bovine bone particulate; autogenous bone graft

STUDY DESIGN:
Who Masked: Participant
Masking Description: the trial is considered a randomized single blind clinical trial due to the following:
  * the participants will be blinded by the technique that will be used during the surgical procedure.
  * the operator will not be blinded for both techniques during the surgical procedure as the two techniques are different.
  * the outcome assessor cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sinus floor elevation And Augmentation using Deproteinized Bovine Bone Particulate. (Active Comparator)
  Interventions: Procedure: maxillary sinus floor elevation using Open Maxillary sinus floor elevation and Augmentation using Deproteinized Bovine Bone Particulate
- Open Maxillary sinus floor elevation and Augmentation using A Mixture of 1:1 Autogenous Bone with De (Experimental)
  Interventions: Procedure: Open Maxillary sinus floor elevation and Augmentation using A Mixture of 1:1 Autogenous Bone with Deproteinized Bovine Bone Particulate

INTERVENTIONS:
Procedure: maxillary sinus floor elevation using Open Maxillary sinus floor elevation and Augmentation using Deproteinized Bovine Bone Particulate — Phase 1: Grafting
  * after administration of Local anesthesia (articaine hydrochloride 68 mg/1.7 ml
    + adrenaline0.017 mg), full-thickness mucoperiosteal flap originating from the mid-crestal area or slightly toward the palate side would be opened.
  * lateral window will be created in the maxillary bone to allow for adequate access to the sinus membrane.
  * The membrane will be carefully elevated using a sinus elevator.
  * bone graft will be placed into the sinus cavity using Autogenous Bone with Deproteinized Bovine Bone Particulate.
  * collagen membrane will be secured in place using resorbable sutures or tacks if necessary.
  Phase 2 (delayed implant placement and core biopsy harvesting 6 Months Postoperative):
  * full thickness mucoperiosteal flap originating from the mid-crestal area or slightly towards palate side would be opened.
  * core biopsy would be harvested using trephine burs from the site of implant placement prior to drilling, to be sent to the Lab for Histological assessment.
  Arms: sinus floor elevation And Augmentation using Deproteinized Bovine Bone Particulate.
Procedure: Open Maxillary sinus floor elevation and Augmentation using A Mixture of 1:1 Autogenous Bone with Deproteinized Bovine Bone Particulate — Phase 1: Grafting
  * After maxillary sinus floor elevation, Mixture of 1:1 Autogenous Bone with Deproteinized Bovine Bone Particulate will be placed in the sinus cavity and secured in place using resorbable sutures or tacks if necessary.
  * Phase 2 (delayed implant placement and core biopsy harvesting 6 Months Postoperative):
    * full thickness mucoperiosteal flap originating from the mid-crestal area or slightly towards palate side would be opened. • core biopsy would be harvested using trephine burs from the site of implant placement prior to drilling, to be sent to the Lab for Histological assessment.
  Arms: Open Maxillary sinus floor elevation and Augmentation using A Mixture of 1:1 Autogenous Bone with De

SUMMARY:
two group of patients with atrophied posterior maxilla that need implant/s placement. one group will be subjected to maxillary sinus floor elevation using 1:1 mixture of autogenous bone and deproteinized bovine bone particulate while the other will be subjected to maxillary sinus floor elevation using deproteinized bovine bone particulate alone.

DETAILED DESCRIPTION:
• Preoperative imaging using CBCT will be performed to assess the anatomy of the maxillary sinus, including the presence of septa, the thickness of the sinus membrane, and the quality and quantity of bone available for grafting and to exlude the presence of any pathosis.

Phase 1 (concerning maxillary sinus floor elevation and Graft placement):

* All surgical procedures will be performed by a single experienced oral surgeon to minimize variability.
* All patients in the two groups would be operated under Local anaesthesia, a full-thickness mucoperiosteal flap originating from the midcrestal area or slightly toward the palate side would be opened.
* A lateral window will be created in the maxillary bone using, The window should be large enough to allow for adequate access to the sinus membrane.
* The Schneiderian membrane will be carefully elevated using a sinus elevator or similar instrument.
* Once the membrane is elevated, Depending on the allocation, graft material will be placed into the sinus cavity either using A mixture of 1:1 Autogenous Bone with Deproteinized Bovine Bone Particulate Versus Deproteinized Bovine Bone Particulate.
* a collagen membrane will be placed over the graft material. The membrane should be trimmed to fit the dimensions of the lateral window and secured in place using resorbable sutures or tacks if necessary.
* The mucoperiosteal flap will be repositioned and secured using sutures.

Phase 2 (delayed implant placement and core biopsy harvesting 6 Months Postoperative):

* A full thickness mucoperiosteal flap originating from the mid-crestal area or slightly towards palate side would be opened for both groups.
* A core biopsy would be harvested from both groups using trephine burs from the site of implant placement prior to drilling, to be sent to the Lab for Histological assessment.

The mucoperiosteal flap will be repositioned and secured using sutures

ELIGIBILITY:
Inclusion Criteria:

* • Patients of both genders requiring implants placement in atrophied posterior maxilla with residual bone height less than 5mm .

  * Patients of age older than 30 years old.
  * Patients with adequate Inter-arch space.
  * Patients who were willing and fully capable to comply with the study protocol.

Exclusion Criteria:

* • Patients suffering from any sinus pathosis

  * Heavy smokers (> than 10 cigarettes a day)
  * Patients with parafunctional habits
  * Patients with uncontrolled systemic diseases.
  * Patients with poor oral hygiene
  * Patients with mental instabilities or psychic patients

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-03-10 (Estimated)

PRIMARY OUTCOMES:
Bone Height Changes | 9 month
  measuring the amount of change in the bone height using cone beam computed tomography in millimeters.

SECONDARY OUTCOMES:
1. Bone Volume Changes | 9 month
  measuring the volumetric changes of bone using CBCT in Cm3

OTHER OUTCOMES:
Percentage of newly formed bone | 9 month
  measuring the percentage of bone area using histomorphometric analysis of decalcified bone sections with hematoxylin and eosin stain using image analyzer computer system
Percentage of Mature Bone | 9 month
  measuring the percentage of mature bone using histomorphometric analysis of decalcified bone sections with masson trichrome stain using image analyzer computer system.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Atef Abdelrasoul, PhD, Study Director — faculty of oral and dental medicine, Cairo university
Locations (1):
- faculty of oral and dental medicine, Cairo university, Cairo, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No